CLINICAL TRIAL: NCT05177328
Title: A Pilot Study to Evaluate the Survival of Transplanted Staphylococcus Hominis A9 on the Skin of Adults With Moderate-to-Severe Atopic Dermatitis (ADRN-13)
Brief Title: Targeted Investigation of Microbiome Elimination
Acronym: TIME-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision to terminate enrollment early was made by the protocol chair and NIAID
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis Research Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ADRN-13
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Masking Description: This is an open-label study, as all participants will receive active and placebo treatment. Participants will receive active treatment on one of their ventral arms and placebo on their contralateral ventral arm. Investigators, all investigational site staff, including those responsible for preparing/administering the investigational product, and all participants in this study will be blinded as to which arm received which treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ShA9 (Experimental): All participants will receive ShA9 active treatment on one of their ventral arms and placebo on their contralateral arm. The assignment of ShA9 and placebo to the dominant and non-dominant arms will be randomized.
  Interventions: Biological: S. hominis A 9 Product; Drug: Placebo

INTERVENTIONS:
Biological: S. hominis A 9 Product — Commensal staph species, phosphate buffered saline, and glycerol.
  Other Names: ShA9
Drug: Placebo — Phosphate buffered saline and glycerol
  Other Names: Placebo for S. hominis A 9 Product

SUMMARY:
The purpose of this study is to examine the pharmacokinetics or survival of new product containing commensal infection fighting bacteria, on the skin of patients with Atopic Dermatitis (AD), after a single application.

DETAILED DESCRIPTION:
This study will enroll a minimum of 20 participants, 18-80 years of age, with moderate-to-severe atopic dermatitis (AD) on their ventral arms. A minimum of 13 participants will have a positive Staphylococcus aureus (S. aureus) colonized lesion on both upper extremities. A minimum of 7 participants will have a negative S. aureus colonized lesion on both upper extremities.

The participant's colonization status will be determined from cultures taken during a pre-treatment phase, approximately 7 days prior to receiving study treatment on Day 0. On Day 0, skin swabs will be collected from lesional and non-lesional sites (at least 21cm^2) on the participant's right and left ventral arms and one non-lesional site on the participant's face. After the skin swab collections, the participant will have ShA9 applied to their right or left ventral arm and placebo applied to their contralateral ventral arm. The assignment of ShA9 and placebo to the dominant and non-dominant arms will be randomized. Additional swabs will be collected 15 minutes, and 1, 2, 4, and 6 hours after the ShA9 and placebo applications on Day 0.

Participants will be asked to return to the clinic 24 hours after receiving their single application and again on Days 3, 10, 17, and 24 for the assessment of adverse events (AEs) and the collection of skin swabs from the identified lesional and non-lesional sites, as needed. After the Day 3 visit, a participant will not be required to complete the Day 10, 17, and 24 visits if their lesional swabs are negative for Coagulase Negative Staphylococcal Species (CoNS).

All randomized participants will complete a final End of Study Phone visit on Day 31 to assess for adverse events and status of their AD.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be able to understand and provide informed consent
2. Meet Atopic Dermatitis Research Network (ADRN) Standard Diagnostic Criteria for active atopic dermatitis (AD)
3. At least 21 cm^2 of lesional and 21 cm^2 of non-lesional skin on both the right and left ventral arms. The required area (lesional or non-lesional) may be one contiguous area or may encompass multiple areas with a total cumulative area of 21 cm^2
4. An Investigator Global Assessment (IGA) score, on the ventral arms of at least moderate severity
5. Body surface area (BSA), as measured by Mostellar BSA Calculator, between 1.26 m^2 and 2.25 m^2
6. If female of child bearing potential, must agree to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraception (e.g. oral contraceptives, intrauterine device [IUD], barrier method with spermicide, or surgically sterilized partner, Depo- Provera, Norplant, NuvaRing, or hormonal implants) for the duration of study participation

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol
2. Pregnant or lactating females
3. Active bacterial, viral, or fungal skin infections
4. Any noticeable breaks or cracks in the skin on the target areas of investigational product application, including severely excoriated skin or skin with open or weeping wounds suggestive of an active infection or increased susceptibility to infection
5. Sensitivity to or difficulty tolerating Dove fragrance-free bar soap, Cetaphil® Lotion, alcohol-based cleaners, glycerol, or soy products
6. Participants with Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
7. Any participant who is immunocompromised (e.g. history of lymphoma, Human Immunodeficiency Virus [HIV]/Acquired Immunodeficiency Syndrome [AIDS], Wiskott-Aldrich Syndrome), has an immune system disorder (e.g. autoimmune disease), or is using a systemic immunosuppressant (e.g. systemic corticosteroids, cyclosporine, methotrexate)
8. Any participant with current malignant disease (with the exception of non-melanoma skin cancer in an area not affected by treatment)
9. Participants with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
10. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
11. Ongoing participation in another investigational trial or use of investigational drugs within 8 weeks, or 5 half-lives (if known), whichever is longer, of the Screening Visit
12. Treatment with non-steroid systemic immunosuppressant within 6 months of the Screening Visit
13. Treatment with Dupilumab within 16 weeks of the Screening Visit
14. Treatment with oral or injectable therapy for AD (excluding oral steroids) within 5 half-lives (if known) or 16 weeks before the Screening Visit, whichever is longer
15. Participants with close contacts (e.g. spouse, children, or members in the same household) that have severe barrier defects or are immunocompromised
16. Use of topical (including steroids and calcineurin inhibitors) AD treatments on the ventral arms or face within 7 days of the Treatment Visit; Use of topical steroids on areas outside of where investigational product is to be applied or swabbing is to be performed may be permitted, per investigator discretion
17. Treatment with prescription moisturizers classified as medical device (e.g., Atopiclair(R), MimyX(R), Epiceram(R), etc.) on the ventral arms or face within 7 days of the Treatment Visit; Use on areas outside of where investigational product is to be applied or swabbing is to be performed is permitted
18. Use of any oral or topical antibiotic within 7 days of the Treatment Visit
19. Participants who have taken a bleach bath within 7 days of the Treatment Visit
20. Use of any oral steroid therapies within 28 days of the Treatment Visit
21. Any phototherapy for skin disease (such as narrow band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + UVA [PUVA]) or regular use (more than 2 visits per week) of a tanning bed within 28 days of the Treatment Visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gallo, M.D., Ph.D., Study Chair — University of California, San Diego: Dermatology Clinical Trials Unit; Tissa Hata, M.D., Study Chair — University of California, San Diego: Dermatology Clinical Trials Unit
Locations (1):
- University of California, San Diego: Dermatology Clinical Trials Unit, La Jolla, California, United States

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was open JUL 2022-OCT 2023. Participants were recruited in person or via phone. Those who met recruitment criteria were invited to an in-clinic Screening Visit where informed consent was given and full eligibility assessed. Those meeting eligibility requirements began a pre-treatment phase for ~7 days before the Day 0 clinic visit.
Pre-assignment Details: 21 participants were enrolled during the recruitment period. Enrolled participants were those who signed informed consent and met all eligibility criteria. 17 of the enrolled participants were randomized and received study therapy. 4 of the enrolled participants discontinued prior to randomization and did not receive study therapy.
Units Other Than Participants: arms
Groups:
- All Randomized Participants: All randomized participants includes participants that were randomized to receive either an application of ShA9 to the dominant ventral arm and placebo to the non-dominant ventral arm, or an application of ShA9 to the non-dominant ventral arm and placebo to the dominant ventral arm.
Period: Overall Study
Arm/Group | All Randomized Participants
Started | 17; 34 arms
Received ShA9 on Dominant Ventral Arm/Placebo on Non-Dominant Ventral Arm | 9; 18 arms
Received ShA9 on Non-Dominant Ventral Arm/Placebo on Dominant Ventral Arm | 8; 16 arms
Completed | 17; 34 arms
Not Completed | 0; 0 arms

BASELINE CHARACTERISTICS:
Population: The safety population includes all participants who were enrolled and received any amount of Staphylococcus hominis A9 (ShA9)/placebo.
Groups:
- Safety Population: The safety population includes all participants who were enrolled and received any amount of Staphylococcus hominis A9 (ShA9)/placebo.
Arm/Group | Safety Population
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17
Staphylococcus aureus (SA) Status [Count of Participants; unit: Participants] — Baseline Staphylococcus aureus (SA) status was defined based on Staphylococcus aureus colony forming unit (CFU) results from samples obtained prior to treatment application during the Treatment Visit (Day 0). Participants were classified as SA Positive if Staphylococcus aureus CFU were greater than or equal to 100 CFU/cm2 for lesional swabs from both arms. Otherwise, participants were classified as SA Negative if Staphylococcus aureus CFU were less than 100 CFU/cm2 for lesional swabs from either arm.
  Participants
    SA Positive | 10
    SA Negative | 7

OUTCOME MEASURES:

1. Primary Outcome: The Duration of ShA9 Survival on the Lesional Ventral Arm Skin of Atopic Dermatitis (AD) Participants Positive for S. Aureus (AD SA+).
Description: Measured as the time needed for coagulase negative staphylococcus species (CoNS) colony-forming unit (CFU) to drop below baseline density measured before application of ShA9 + 100 CFU/cm2 (time to CoNS elimination). Baseline CoNS density was defined as the CoNS (CFU/cm2) result from the sample taken prior to treatment application during the Treatment Visit (Day 0). The primary endpoint was assessed based on samples from lesional skin from the arm (left or right) that received active treatment (ShA9) among SA+ participants. The event is CoNS elimination. Participants who did not experience CoNS elimination were right-censored. The median survival time (hours) was estimated using Kaplan Meier techniques. The 95% confidence interval for median survival time was estimated based on a log-log transformation of the survivor function.
Time Frame: Day 0 to Day 24
Measure: Median (95% Confidence Interval); unit: Hours
Groups:
- mITT, SA+ Participants: The modified intent-to-treat (mITT) population includes all participants who were enrolled and received any amount of study product (ShA9 or placebo). The analysis of the primary endpoint is subset to the mITT participants who were SA+ at baseline [based on samples obtained prior to treatment application during the Treatment Visit (Day 0)]. Out of the 10 participants who were analyzed, the number of participants who were censored equals 0.
Arm/Group | mITT, SA+ Participants
Number analyzed (Participants) | 10
Hours | 37.0 [0.25 to 240.00]

2. Secondary Outcome: The Duration of ShA9 Survival on the Non-lesional Ventral Arm Skin of Atopic Dermatitis (AD) Participants Positive for S. Aureus (AD SA+).
Description: Measured as the time needed for coagulase negative staphylococcus species (CoNS) colony-forming unit (CFU) to drop below baseline density measured before application of ShA9 + 100 CFU/cm2 (time to CoNS elimination). Baseline CoNS density was defined as the CoNS (CFU/cm2) result from the sample taken prior to treatment application during the Treatment Visit (Day 0). This secondary endpoint was assessed based on samples from non-lesional skin from the arm (left or right) that received active treatment (ShA9) among SA+ participants. The event is CoNS elimination. Participants who did not experience CoNS elimination were right-censored. The median survival time (hours) was estimated using Kaplan Meier techniques. The 95% confidence interval for median survival time was estimated based on a log-log transformation of the survivor function.
Time Frame: Day 0 to Day 24
Measure: Median (95% Confidence Interval); unit: Hours
Groups:
- mITT, SA+ Participants: The modified intent-to-treat (mITT) population includes all participants who were enrolled and received any amount of study product (ShA9 or placebo). The analysis of the primary endpoint is subset to the mITT participants who were SA+ at baseline [based on samples obtained prior to treatment application during the Treatment Visit (Day 0)]. Out of the 10 participants who were analyzed, the number of participants who were censored equals 1.
Arm/Group | mITT, SA+ Participants
Number analyzed (Participants) | 10
Hours | 6.0 [0.25 to 24.00]

3. Secondary Outcome: The Count of Serious Treatment-emergent Adverse Events Per Participant.
Description: For this study, an adverse event included any untoward or unfavorable medical occurrence associated with the study treatment regimen or study mandated procedures. An adverse event was considered 'serious' if, in the view of the investigator or Sponsor, it resulted in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 0 to Day 31
Measure: Mean (Standard Deviation); unit: Serious TEAEs per participant
Arm/Group | Safety Population
Number analyzed (Participants) | 17
Serious TEAEs per participant | 0 (0)

4. Secondary Outcome: The Count of Non-serious Treatment-emergent Adverse Events Per Participant.
Description: For this study, an adverse event included any untoward or unfavorable medical occurrence associated with the study treatment regimen or study mandated procedures. An adverse event was considered 'non-serious' if it did not result in any of the serious defined outcomes.
Time Frame: Day 0 to Day 31
Measure: Mean (Standard Deviation); unit: Non-serious TEAEs per participant
Arm/Group | Safety Population
Number analyzed (Participants) | 17
Non-serious TEAEs per participant | 0.24 (0.752)

ADVERSE EVENTS:
Time Frame: Screening through Day 31
Description: Adverse events (AEs) were collected from Screening-Day 31. AEs included any untoward/unfavorable medical occurrence associated with study treatment or study mandated procedures. AEs are reported for enrolled subjects. Treatment-emergent AEs were summarized by involvement of ShA9 or placebo-treated arm. AEs involving both arms were counted in both arm summaries. AEs involving both arms and other body parts were also counted as systemic. AEs occurring prior to treatment were considered systemic.
Groups:
- ShA9-Treated Ventral Arm: Treatment-emergent adverse events involving the ShA9-treated ventral arm among participants included in the safety population.
- Placebo-Treated Ventral Arm: Treatment-emergent adverse events involving the placebo-treated ventral arm among participants included in the safety population.
- Systemic: Systemic adverse events among all enrolled participants.
- Overall: All adverse events for enrolled participants.
Arm/Group | ShA9-Treated Ventral Arm | Placebo-Treated Ventral Arm | Systemic | Overall
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 2/17 | 2/17 | 3/21 | 3/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ShA9-Treated Ventral Arm (N=17) | Placebo-Treated Ventral Arm (N=17) | Systemic (N=21) | Overall (N=21)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bipolar II disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT05177328/Prot_001.pdf
  • Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT05177328/SAP_002.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT05177328/ICF_000.pdf